CLINICAL TRIAL: NCT03417843
Title: A Prospective, Open Label Study: Safety and Efficacy of a New Ablation Catheter RFA (Radiofrequency Under EUS) Developed by TAEWOONG Company for the Treatment of Pancreatic Premalignant and Early Malignant Cyctic Lesions.
Brief Title: Safety and Efficacy of an Ablation Catheter for the Treatment of Pancreatic Premalignant Cyctic Lesions.
Acronym: yes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Stanislav Bezobchuk, senior of gasroenterology, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0090-17-EMC
Record Dates: First submitted 2018-01-17; First posted 2018-01-31 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Cancer; Pancreatic Neuroendocrine Tumor; Pancreatic Cyst; Pancreatic Cancer Stage
Keywords: ablation catheter; pancreatic premalignant and early malignant cystic lesion
MeSH Terms: conditions — Pancreatic Neoplasms; Adenoma, Islet Cell; Pancreatic Cyst

STUDY DESIGN:
Intervention Model Description: A Prospective, open- label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUSRA RF electrode (Experimental): new ablation catheter RFA (RADIOFREQUENCY under EUS), developed by TAEWOONG company for the treatment of pancreatic premalignant and early malignant cystic lesion.
  Interventions: Device: EUSRA RF electrode

INTERVENTIONS:
Device: EUSRA RF electrode — At the tip of the needle there is a probe that releases the peripheral energy in a continuous and continuous manner. The method is a long 50W power release for 10 seconds or 40W until white bubbles appear in a sonographic image.
  Materials that come into contact with the body: electrode and grounding surfaces

SUMMARY:
This study aims to evaluate the safety and efficacy of new ablation catheter developed by MEDICAL TAEWOONG for the treatment of pancreatic premalignant and early malignant cystic lesion. The ablation is performed using EUSRA needle and radiofrequncy waves under ultrasound imaging. The method will be exaimened on patients who are candidates for surgical intervention and to examine the ability of the method to serve as an alternative to surgical intervention.

DETAILED DESCRIPTION:
In recent years, local and non-invasive intervention methods have been attempted to eliminate or at least reduce the growth of pancreatic lesions. Over the past two years there has been considerable but not successful experience in ablation (burning) of lesions by direct alcohol injection and / or other drugs into the cyst through the EUS. To date, treatment has been performed in three groups of patients in a clinical trial and has shown clinical success from 33% to 70%. However, it should be noted that there is a large incidence of treatment failure and also complications such as pancreatitis.

An interesting alternative to surgical intervention is the local destruction of the cyst by radio waves ENDOSCOPIC RADIOFREQUENCY (RF). This is a familiar local method that works by releasing heat that causes necrosis and disappearance of the lesion.High efficacy and high safety profile were reported for this method; 90% of the cases showed disappearance of of metaplasia by the follow-up of 5 years and 80% disappearance of dysplasia (both early and advanced) followed by two and a half years.

In addition, in recent years EMCISION has developed a catheter called ENDO HBP HABIB. It is a thin RF probe that can be inserted through work channels of all types of endoscopes and cholangioscopes. The depth of the penetration of heat and energy intensity is in accordance with the resistance of the tissue being treated, and the device operates under the computerized control of an ultrasound device with high resolution. This method showed success in short-term follow-up in preliminary research.The technical difficulty of this therapeutic method is related to the limitation of the ability to position itself precisely by inserting the catheter through the EUS needle.In order to overcome the difficulty of operating HABIB PROBE, MEDICAL TAEWOONG, recognized worldwide and Israel as an advanced endoscopic equipment company, developed in cooperation with STARMED an RF needle called EUSRA, which works in conjunction with a VIVO COMBO generator. The function of the generator is to provide up to 200 watts of energy to activate the electrode. The needle can be directly inserted into the pancreas lesion while controlling EUS. At the tip of the needle is a probe that releases the energy at 50W for 10 seconds or 40W until the white bubbles appear in a sonographic image.In recent years, two cases of successful treatment have been reported. In both cases, treatment of neuroendocrine cancer showed good initial results. The first study was performed on a 76-year-old patient with a neuroendocrine tumor.CT performed about one month after the procedure showed complete disappearance of the lesion without any complications. The second study was performed in six patients with an average age of 62. The average diameter of lesion was 3.8 cm. The procedure was successful when two patients felt abdominal pain followed. There were no bleeding events and pancreatitis.This year, a multicenter study was conducted in France in patients with neuroendocrine tumors and cystic lesions in the pancreas, testing the safety and initial efficacy of the method and monitoring for up to 12 months. The study was conducted in a group of 30 patients.In 6 patients with endocrine tumors there was complete disappearance of the lesions, in 3 patients there was a decrease in the diameter of the lesions by more than 50% and in one patient the treatment failed. In 7 of 8 patients with cystic tumors, walled nadies disappeared and in 5 out of 10 patients cystic tumors disappeared. Prophylactic treatment of antibiotics and NSAIDs (anti-inflammatory drugs) and empty the cyst fluid before the procedure led to a dramatic reduction in complications (3.5%). Three patients experienced mild abdominal pain without signs of inflammation successfully treated with paracetamol. (study not yet published).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85

  • Patients who agreed to join study and signed an informed consent letter
* Patients with IPMN pancreas cystic tumor with a diameter greater than 30 mm and with secondary branches.

  * Patients with a tissue component within the cystic lesion
  * Patients with atypical cells in cytology, regardless of the size of the lesion and regardless of the contents of the cyst
  * Patients with a lesion of less than 30 mm diameter showing rapid changes in size (15 mm increments followed by 6 months)
  * Patients with a consistent increase in CEA level within the cyst.
  * Patients with cystinus cystadenoma of any size with suspicious signs such as thickening of the cyst wall, calcification of the cyst wall, irregularity of the cyst wall, tissue content within the cyst, the presence of atypical cells within the cyst in cytology.
  * Symptomatic patients (pain defined as related to the lesion)
  * Asymptomatic patients with a normal cyst greater than 40 mm in diameter.
  * Patients referred for surgical treatment (after the multidisciplinary committee (gastroenterologists, surgeons and pathologists / cytologists) has approved the diagnosis and indication of therapeutic intervention (as is customary) but not suitable for surgery due to high risk of anesthesia (ASAIV) or severe anatomy due to repeat surgery or patients who do not agree to undergo surgical intervention (these are most patients)
  * Patients with low anesthetic risk: ASA 1-3.
  * Women who are not pregnant during recruitment, and women of childbearing age who take birth control during the study.

Exclusion Criteria:

* Patients with clear evidence of invasive tumor development within the lesion (both candidates and not candidates for continued surgical treatment).
* Patients with severe coagulation disorders (PT, elongated PTT)
* Patients with platelet counts less than 75000
* Patients taking anticoagulants that can not be stopped temporarily
* Patients with pacemakers
* Patients with dilatation pages
* Patients who take clopidogrel in situations that do not allow temporary cessation of the drug.
* Patients with hight anesthetic risk(ASA4 group).
* Patients belonging to groups: pregnant women, nursing patients, and demineral patients.
* Women of childbearing age who do not take birth control.
* Patients who are unable to express informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse and serious adverse events | up to one month post-procedure
  The number of subjects with post EUS-RFA-related adverse events including:
  Fever >38C (will be measured in celcius)
Incidence of adverse and serious adverse events | up to 72 hours post-procedure
  The number of subjects with post EUS-RFA-related adverse events including:
  Pancreatitis as measured by an increase of at least 3 times in serum amylase (units/liter) in the initial 72 hours post-procedure
Incidence of adverse and serious adverse events | up to 72 hours post-procedure
  The number of subjects with post EUS-RFA-related adverse events including:
  Hemorrhage as measured by need for transfusion of packed red blood cells
Incidence of adverse and serious adverse events | up to 72 hours post-procedure
  The number of subjects with post EUS-RFA-related adverse events including:
  Perforation as confirmed by abdominal CT
Incidence of adverse and serious adverse events | up to 12 months post-procedure
  The number of subjects with post EUS-RFA-related adverse events including:
  Mortality

SECONDARY OUTCOMES:
Absolute disappearance incidence or reduction in lesion size | up to 12 months post-procedure (3, 6 and 12 months post-procedure)
  Direct measuring of lesion diameter and area (in milimeter and milimeter^2 respectively) during the 12-month blind follow-up by EUS, CT and MRI .
Absolute disappearance incidence or reduction in lesion size | up to 12 months post-procedure (3, 6 and 12 months post-procedure)
  disappearance of mural nodule inside cyst follow-up by EUS, CT and MRI .
Technical efficiency of the method | during the procedure
  To examine the technical efficiency of the method by estimating the frequency of success in performing the operation according to the protocol, without any mishaps and deviations from the original protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Bezobchuk, doctor, Principal Investigator — HaEmek Medical Center, Israel

IPD SHARING:
Plan to Share IPD: Yes
IPD for study protocol will made avilable
Supporting Information: Study Protocol
Time Frame: 12 months since study completion
Access Criteria: data access requests will be reviewed by an external independent review panel. Requestors will be requested to sign a data acess agreement

REFERENCES:
- [Background] Hammel P. [Incidental pancreatic tumors: diagnosis and management]. Gastroenterol Clin Biol. 2002 Aug-Sep;26(8-9):700-8. No abstract available. French. PMID 12434071
- [Background] Brugge WR, Lewandrowski K, Lee-Lewandrowski E, Centeno BA, Szydlo T, Regan S, del Castillo CF, Warshaw AL. Diagnosis of pancreatic cystic neoplasms: a report of the cooperative pancreatic cyst study. Gastroenterology. 2004 May;126(5):1330-6. doi: 10.1053/j.gastro.2004.02.013. PMID 15131794
- [Background] Okabayashi T, Kobayashi M, Nishimori I, Sugimoto T, Namikawa T, Okamoto K, Okamoto N, Kosaki T, Onishi S, Araki K. Clinicopathological features and medical management of intraductal papillary mucinous neoplasms. J Gastroenterol Hepatol. 2006 Feb;21(2):462-7. doi: 10.1111/j.1440-1746.2005.03958.x. PMID 16509876
- [Background] Matsumoto T, Aramaki M, Yada K, Hirano S, Himeno Y, Shibata K, Kawano K, Kitano S. Optimal management of the branch duct type intraductal papillary mucinous neoplasms of the pancreas. J Clin Gastroenterol. 2003 Mar;36(3):261-5. doi: 10.1097/00004836-200303000-00014. PMID 12590239
- [Background] Gan SI, Thompson CC, Lauwers GY, Bounds BC, Brugge WR. Ethanol lavage of pancreatic cystic lesions: initial pilot study. Gastrointest Endosc. 2005 May;61(6):746-52. doi: 10.1016/s0016-5107(05)00320-2. PMID 15855986
- [Background] Oh HC, Seo DW, Lee TY, Kim JY, Lee SS, Lee SK, Kim MH. New treatment for cystic tumors of the pancreas: EUS-guided ethanol lavage with paclitaxel injection. Gastrointest Endosc. 2008 Apr;67(4):636-42. doi: 10.1016/j.gie.2007.09.038. Epub 2008 Feb 11. PMID 18262182
- [Background] DeWitt J, McGreevy K, Schmidt CM, Brugge WR. EUS-guided ethanol versus saline solution lavage for pancreatic cysts: a randomized, double-blind study. Gastrointest Endosc. 2009 Oct;70(4):710-23. doi: 10.1016/j.gie.2009.03.1173. Epub 2009 Jul 4. PMID 19577745
- [Background] Cho YK, Kim JK, Kim MY, Rhim H, Han JK. Systematic review of randomized trials for hepatocellular carcinoma treated with percutaneous ablation therapies. Hepatology. 2009 Feb;49(2):453-9. doi: 10.1002/hep.22648. PMID 19065676
- [Background] Fleischer DE, Overholt BF, Sharma VK, Reymunde A, Kimmey MB, Chuttani R, Chang KJ, Muthasamy R, Lightdale CJ, Santiago N, Pleskow DK, Dean PJ, Wang KK. Endoscopic radiofrequency ablation for Barrett's esophagus: 5-year outcomes from a prospective multicenter trial. Endoscopy. 2010 Oct;42(10):781-9. doi: 10.1055/s-0030-1255779. Epub 2010 Sep 20. PMID 20857372
- [Background] Shaheen NJ, Sharma P, Overholt BF, Wolfsen HC, Sampliner RE, Wang KK, Galanko JA, Bronner MP, Goldblum JR, Bennett AE, Jobe BA, Eisen GM, Fennerty MB, Hunter JG, Fleischer DE, Sharma VK, Hawes RH, Hoffman BJ, Rothstein RI, Gordon SR, Mashimo H, Chang KJ, Muthusamy VR, Edmundowicz SA, Spechler SJ, Siddiqui AA, Souza RF, Infantolino A, Falk GW, Kimmey MB, Madanick RD, Chak A, Lightdale CJ. Radiofrequency ablation in Barrett's esophagus with dysplasia. N Engl J Med. 2009 May 28;360(22):2277-88. doi: 10.1056/NEJMoa0808145. PMID 19474425
- [Background] Monga A, Gupta R, Ramchandani M, Rao GV, Santosh D, Reddy DN. Endoscopic radiofrequency ablation of cholangiocarcinoma: new palliative treatment modality (with videos). Gastrointest Endosc. 2011 Oct;74(4):935-7. doi: 10.1016/j.gie.2010.10.018. Epub 2010 Dec 18. No abstract available. PMID 21168839
- [Background] Steel AW, Postgate AJ, Khorsandi S, Nicholls J, Jiao L, Vlavianos P, Habib N, Westaby D. Endoscopically applied radiofrequency ablation appears to be safe in the treatment of malignant biliary obstruction. Gastrointest Endosc. 2011 Jan;73(1):149-53. doi: 10.1016/j.gie.2010.09.031. PMID 21184881
- [Background] Dolak W, Schreiber F, Schwaighofer H, Gschwantler M, Plieschnegger W, Ziachehabi A, Mayer A, Kramer L, Kopecky A, Schrutka-Kolbl C, Wolkersdorfer G, Madl C, Berr F, Trauner M, Puspok A; Austrian Biliary RFA Study Group. Endoscopic radiofrequency ablation for malignant biliary obstruction: a nationwide retrospective study of 84 consecutive applications. Surg Endosc. 2014 Mar;28(3):854-60. doi: 10.1007/s00464-013-3232-9. Epub 2013 Oct 3. PMID 24196547
- [Background] Prat F, Lafon C, De Lima DM, Theilliere Y, Fritsch J, Pelletier G, Buffet C, Cathignol D. Endoscopic treatment of cholangiocarcinoma and carcinoma of the duodenal papilla by intraductal high-intensity US: Results of a pilot study. Gastrointest Endosc. 2002 Dec;56(6):909-15. doi: 10.1067/mge.2002.129872. PMID 12447312
- [Background] Itoi T, Isayama H, Sofuni A, Itokawa F, Tamura M, Watanabe Y, Moriyasu F, Kahaleh M, Habib N, Nagao T, Yokoyama T, Kasuya K, Kawakami H. Evaluation of effects of a novel endoscopically applied radiofrequency ablation biliary catheter using an ex-vivo pig liver. J Hepatobiliary Pancreat Sci. 2012 Sep;19(5):543-7. doi: 10.1007/s00534-011-0465-7. PMID 22038500
- [Background] Zacharoulis D, Lazoura O, Rountas C, Katsimboulas M, Mantzianas G, Tzovaras G, Habib N. Experimental animal study of a novel radiofrequency endovascular occlusion device. Am J Surg. 2011 Jul;202(1):103-9. doi: 10.1016/j.amjsurg.2010.08.031. PMID 21741521
- [Background] Kim HJ, Seo DW, Hassanuddin A, Kim SH, Chae HJ, Jang JW, Park DH, Lee SS, Lee SK, Kim MH. EUS-guided radiofrequency ablation of the porcine pancreas. Gastrointest Endosc. 2012 Nov;76(5):1039-43. doi: 10.1016/j.gie.2012.07.015. PMID 23078928
- [Background] Armellini E, Crino SF, Ballare M, Occhipinti P. Endoscopic ultrasound-guided radiofrequency ablation of a pancreatic neuroendocrine tumor. Endoscopy. 2015;47 Suppl 1 UCTN:E600-1. doi: 10.1055/s-0034-1393677. Epub 2015 Dec 15. No abstract available. PMID 26671543
- [Background] Song TJ, Seo DW, Lakhtakia S, Reddy N, Oh DW, Park DH, Lee SS, Lee SK, Kim MH. Initial experience of EUS-guided radiofrequency ablation of unresectable pancreatic cancer. Gastrointest Endosc. 2016 Feb;83(2):440-3. doi: 10.1016/j.gie.2015.08.048. Epub 2015 Sep 4. PMID 26344883
- [Background] Preliminary data of first RFA results of Multicentre study in France (not published). Oral presentation RFA course , Marseille 05.2017.